CLINICAL TRIAL: NCT05334550
Title: Effectiveness of Home Based Early Intervention of Extremely Premature Infant by Parent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-02-28
Record Dates: First submitted 2022-03-02; First posted 2022-04-19 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Preterm; Extreme Prematurity; Early Intervention; Developmental Delay; Motor Outcome; Home Exercise; Parents
MeSH Terms: conditions — Premature Birth; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Allocated to intervention group through randomization process.
  Interventions: Other: Home Based Early Intervention by Parent
- Control group (No Intervention): Allocated to control group through randomization process.

INTERVENTIONS:
Other: Home Based Early Intervention by Parent — Through a video communication program called ZOOM, the parents of intervention group are educated once every two weeks for three months. Parent education consists of a program developed by our pediatric rehabilitation therapist to help premature infants develop motor skills. Parents provide daily exercise training to their children as educated.
  Arms: Intervention group

SUMMARY:
This study is to prove the effectiveness of home based early intervention of extremely premature infant by Parent.

DETAILED DESCRIPTION:
The perpose of this study to prove the significance of the hypothesis that there will be a significant improvement in motor development when remote tele-rehabilitation treatment is performed for extremely premature infants. The investigators plan to recruit subjects who meet the inclusion criteria and do not meet the exclusion criteria from among extremely premature infants born at Samsung Hospital, Seoul, Korea, whose gestational age is from 23 weeks to 28 weeks. The target number of n is 110, 55 per group. After randomization into an intervention group and a control group, the intervention group get the intervention starting at 0 months of correctional age and runs for 3 months. In both groups, motor outcomes are measured at the time of enrollment, at 3 months of correction age, 6 months of correction age and 12 months of correction age

ELIGIBILITY:
Inclusion Criteria:

* Extreme premature baby (gestationl age 23~28 weeks)
* Corrected age under one month at the time of enroll of this study
* Children of those who voluntarily decided to participate after hearing detailed explanations about this study and gave their written consent.
* Children whose parents are Korean

Exclusion Criteria:

* Congenital anomalies in the central nervous system
* Hereditary diseases
* Chromosomal abnormalities (Down syndrome, etc.)
* Stage 3 or more intraventricular hemorrhage
* If surgery was performed for hydrocephalus
* Leukomalacia confirmed by ultrasound examination (not applicable to increase in white matter shading)
* Neonatal asphyxia
* Other central nervous system diseases
* If taking medications for convulsions or epilepsy
* Metabolic disease
* In the case of premature infants undergoing surgery for retinal disease
* Hearing loss
* In case of surgery due to complex congenital anomaly or planned operation (not excluded if surgery is not required)
* In case of oxygen dependence due to lung disease in premature infants
* Musculoskeletal disorders (hip dislocation, polyarthrosis, etc.)
* Neuromuscular disease, etc.
* Those whose family has social problems
* Those whose parents cannot participate in this study
* Those who have other serious complications that cannot proceed with the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-06-02 (Estimated); Primary Completion 2023-03-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Test of infant motor performance at 3 months | around the start of intervention(up to 1 week), 3 months after the start of intervetion
  The Test of infant motor performance (TIMP) is conducted on infants under 4 months of age to perform functions in daily life. It is performed to evaluate the selective control of postures and movements that infants need in daily life, and takes an average of 25-35 minutes. The TIMP was developed to 1) identify infants with delayed motor development, 2) differentiate between infants with varying degrees of risk for measurement outcomes, and 3) measure changes due to interventions. Because it can be used in both early intervention programs, it can aid in communication between parents and health care providers in a variety of settings. The range of test score is from 0 to 142. The higher score means the better motor performance.

SECONDARY OUTCOMES:
Change from baseline Edinburgh postnatal depression scale at 3 months | around the start of intervention(up to 1 week), 3 months after the start of intervetion
  Edinburgh postnatal depression scale is a 10-item scale for screening for maternal depression. Each item is scored from 0 to 3; the higher score indicates the possibility of depressed status. Total score is from 0 to 30. A score of 13 or higher indicates a possible postpartum depression. It has been validated by several studies confirming that EPDS is a reliable and sensitive indicator of depression.
Alberta infant motor scale | 6 months and 12 months after the start of intervetion
  Alberta infant motor scale is a validated and reliable observational tool for use in infants from full term to 18 months of age. Alberta infant motor scale can evaluate the qualitative aspects of movement and sensitively measure the change in infant's motor performance. Assessment of Alberta infant motor scale is scored based on the number of gross motor postures and movements the infant has demonstrated while prone, supine, and sitting or standing. The range of scores of each item are as followed; prone is from 0 to 21, supine is from 0 to 9, sitting is from 0 to 12, standing is from 0 to 16. The range of total score is from 0 to 58. The higher score means the better motor performance. The evaluation score can be converted to a percentile rank that can be compared with the percentile rank of a standard age-matched infant sample.
Peabody Developmental Motor Scales 2nd edition | 12 months after the start of intervetion
  Peabody Developmental Motor Scales 2nd edition evaluates both fine motor and macromotor function. It can be evaluated from newborn to 5 years old. It consists of six subtests: reflex, stationary, locomotion, object manipulation, grasping, and visual motor integration. Range of score of each items are as followed; reflex is from 0 to 16, stationary is from 0 to 60, locomotion is from 0 to 198, objective manipulation is from 0 to 48, grasping is from 0 to 26, visual-motor integration is from 0 to 72. The summation of scores is converted into age-matched percentile that can be ranked. The higher scores is matched to better ranked percentile. Peabody Developmental Motor Scales 2nd edition is a test whose reliability and validity have been verified in various conditions such as autism, cerebral palsy, and premature infants.

CONTACTS AND LOCATIONS:
Overall Officials: Kwon Jeong-Yi, PhD, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 통계청, 『2019년 출생통계(확정), 국가승인통계 제10103호 출생통계』
- [Background] McIntire DD, Leveno KJ. Neonatal mortality and morbidity rates in late preterm births compared with births at term. Obstet Gynecol. 2008 Jan;111(1):35-41. doi: 10.1097/01.AOG.0000297311.33046.73. PMID 18165390
- [Background] Morgan AM, Koch V, Lee V, Aldag J. Neonatal neurobehavioral examination. A new instrument for quantitative analysis of neonatal neurological status. Phys Ther. 1988 Sep;68(9):1352-8. doi: 10.1093/ptj/68.9.1352. PMID 3420169
- [Background] Piper MC, Darrah J. Motor Assessment of the Developing Infant. Philadelphia: WB Saunders; 1994.
- [Background] Aita M, De Clifford Faugere G, Lavallee A, Feeley N, Stremler R, Rioux E, Proulx MH. Effectiveness of interventions on early neurodevelopment of preterm infants: a systematic review and meta-analysis. BMC Pediatr. 2021 Apr 29;21(1):210. doi: 10.1186/s12887-021-02559-6. PMID 33926417
- [Background] Fernández Rego Francisco Javier, Gómez Conesa Antonia, Pérez López Julio, Efficacy of Early Physiotherapy Intervention in Preterm Infant Motor Development- A Systematic Review-, Journal of Physical Therapy Science, 2012, Volume 24, Issue 9, Pages 933-940, Released December 01, 2012, Online ISSN 2187-5626, Print ISSN 0915-5287
- [Background] Puthussery S, Chutiyami M, Tseng PC, Kilby L, Kapadia J. Effectiveness of early intervention programs for parents of preterm infants: a meta-review of systematic reviews. BMC Pediatr. 2018 Jul 9;18(1):223. doi: 10.1186/s12887-018-1205-9. PMID 29986683
- [Background] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166
- [Background] 배영임, 신혜리. 코로나19, 언택트 사회를 가속화하다. 이슈&진단 . (2020): 1-26.
- [Background] Campbell SK, Wright BD, Linacre JM. Development of a functional movement scale for infants. J Appl Meas. 2002;3(2):190-204. PMID 12011500
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Boyce P, Stubbs J, Todd A. The Edinburgh Postnatal Depression Scale: validation for an Australian sample. Aust N Z J Psychiatry. 1993 Sep;27(3):472-6. doi: 10.3109/00048679309075805. PMID 8250792
- [Background] Milgrom J, Ericksen J, Negri L, Gemmill AW. Screening for postnatal depression in routine primary care: properties of the Edinburgh Postnatal Depression Scale in an Australian sample. Aust N Z J Psychiatry. 2005 Sep;39(9):833-9. doi: 10.1080/j.1440-1614.2005.01660.x. PMID 16168042
- [Background] Piper MC, Pinnell LE, Darrah J, Maguire T, Byrne PJ. Construction and validation of the Alberta Infant Motor Scale (AIMS). Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S46-50. PMID 1468050
- [Background] Martin T. Stein, Meghan Korey Lukasik, Chapter 79 - DEVELOPMENTAL SCREENING AND ASSESSMENT: INFANTS, TODDLERS, AND PRESCHOOLERS, Editor(s): William B. Carey, Allen C. Crocker, William L. Coleman, Ellen Roy Elias, Heidi M. Feldman, Developmental-Behavioral Pediatrics (Fourth Edition), W.B. Saunders, 2009, Pages 785-796,
- [Background] Fan J, Wang J, Zhang X, He R, He S, Yang M, Shen Y, Tao X, Zhou M, Gao X, Hu L. A home-based, post-discharge early intervention program promotes motor development and physical growth in the early preterm infants: a prospective, randomized controlled trial. BMC Pediatr. 2021 Apr 7;21(1):162. doi: 10.1186/s12887-021-02627-x. PMID 33827496
- [Background] Holloway JM, Long TM, Biasini F. Relationships Between Gross Motor Skills and Social Function in Young Boys With Autism Spectrum Disorder. Pediatr Phys Ther. 2018 Jul;30(3):184-190. doi: 10.1097/PEP.0000000000000505. PMID 29727358
- [Background] Clutterbuck GL, Auld ML, Johnston LM. High-level motor skills assessment for ambulant children with cerebral palsy: a systematic review and decision tree. Dev Med Child Neurol. 2020 Jun;62(6):693-699. doi: 10.1111/dmcn.14524. Epub 2020 Apr 1. PMID 32237147
- [Background] Tavasoli A, Azimi P, Montazari A. Reliability and validity of the Peabody Developmental Motor Scales-second edition for assessing motor development of low birth weight preterm infants. Pediatr Neurol. 2014 Oct;51(4):522-6. doi: 10.1016/j.pediatrneurol.2014.06.010. Epub 2014 Jun 24. PMID 25266615
- [Background] Wang M, Mei H, Liu C, Zhang Y, Huixian LI, Yan F. Application of the Peabody developmental motor scale in the assessment of neurodevelopmental disorders in premature infants. Chinese Pediatric Emergency Medicine. 2017 Jan 1;24(10):760-3.